CLINICAL TRIAL: NCT00163618
Title: Multicenter Phase IV Study to Investigate the Seropersistence of TBE Virus Antibodies Approx. 3 Years After a Booster Vaccination With FSME-IMMUN 0.25 mL JUNIOR in Children
Brief Title: Study to Investigate the Seropersistence of TBE Virus Antibodies Approx. 3 Years After a Booster Vaccination With FSME-IMMUN 0.25 mL JUNIOR in Children
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 700501
Record Dates: First submitted 2005-09-08; First posted 2005-09-14 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
Keywords: tick-borne encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Formaldehyde inactivated, sucrose gradient purified TBE virus antigen, strain Neudörfl

SUMMARY:
The objective of this study is to assess the TBE antibody persistence approximately three years after administration of a TBE booster vaccination with FSME-IMMUN 0.25 ml Junior in children who received either 0.25 mL or 0.5 mL TicoVac for their primary vaccination series in Study 146A.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children who participated in Study 146A if:
* they and/or their parents/legal guardians understand the nature of the study and agree to its provisions
* written informed consent is available from the child (according to age and capacity of understanding) and the parents/legal guardians
* they received the complete 3-immunization primary vaccination series with either 0.5 ml or 0.25 ml TicoVac in Study 146A
* they received FSME-IMMUN 0.25 ml Junior for their first booster vaccination approximately 3 to 4 years after their third vaccination in Study IMAG-146A

Exclusion Criteria:

* Subjects who received any further TBE vaccination since their first TBE booster vaccination
* Subjects with a history of infection with, or vaccination against, other flaviviruses (e.g. dengue fever, yellow fever and/or japanese B encephalitis virus) since their third vaccination in Study 146A
* Subjects who have suffered from a disease (e.g. autoimmune disease) or have undergone a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions within 30 days before and after their first TBE booster vaccination
* Subjects who have been known to be HIV positive (a special HIV test is not required for the purpose of the study) since their third vaccination in Study 146A
* Subjects who have received a blood transfusion or immunoglobulins within 30 days of study entry

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2005-06; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (4):
- Austria (4):
  - Bahnhofstraße 9, Hermagor
  - Freistädter Strasse 290, Linz
  - Conrad-von-Hoetzendorf-Strasse, Voitsberg
  - Grieskirchner Strasse 17, Wels